

#### **Research title:**

Comparing the Effect of Early Childhood Caries Treatment Procedures Under General and Local anesthesia on the Quality of Life of Young Children

# **Document Type:** Informed Consent Form

**NCT Number:** Not yet assigned

## **Document Date:** 01- 01- 2021

## Principle Investigator: Mohammad Alwadaani

# **Sponsor:** Nill

IRB Approval Number: FBGRP-2021-562-421-415

#### **Participating Site:**

Riyadh Elm University, Riyadh, KSA



You are requested to participate in research that will be supervised by Dr.Mohammad Alwadaani in Riyadh Elm University. This study is about Comparing the effect of ECC treatment procedures under general and local anesthesia on the OHRQoL of young children.

Your participation is voluntary and you have the right not to accept filling this survey without giving any reason and this will not affect your current or future medical care in REU hospitals.

You don't have to sign this information sheet only you can choose to agree/disagree; your acceptance to complete the survey will be interpreted as your informed consent to participate. Your responses will be kept anonymous. If you have any questions about the research, Please contact (Dr.Mohammad Alwadaani - Riyadh city- Mobile:0550226711)

| ( ) Agree to participate ( ) Disagree to participate | ( ) Agree to participate | () Disagree to participat |
|---|---|---|
|---|---|---|

| Age of child: |
|---|
| Gender: |
| Location: ( ) Urban ( ) Rural |
| Father's education: ( ) Elementary school ( ) Intermediate school ( ) Secondary school ( ) University |
| Mother's education: ( ) Elementary school ( ) Intermediate school ( ) Secondary school ( ) University |
| Father working: Yes NO |
| Mother working: Yes NO |
| Family income (monthly): () Low (Below 10,000 SAR) () Moderate (Between 10,000 SAR to 30,000 SAR) () HIGH (Above 30,000 SAR) |

| Impacts | Never | Hardly ever | Occasionally | Often | Very often | I don't know |
|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 |
| Child impact | | | | | | |
| 1-Dental pain | | | | | | |
| 2-Difficulty drinking | | | | | | |
| 3-Diffculty eating | | | | | | |
| 4-Diffculty pronouncing word | | | | | | |
| 5-Missed preschool or school | | | | | | |
| 6-Trouble sleeping | | | | | | |
| 7-Irritable or frustrated | | | | | | |
| 8-Avoid smiling or laughing | | | | | | |
| 9-Avoid talking | | | | | | |
| Family impact | | | | | | |
| 10-Been upset | | | | | | |
| 11-Felt guilty | | | | | | |
| 12-Time off from work | | | | | | |
| 13-Financial impact | | | | | | |

<sup>&#</sup>x27;How would you rate your child's current OH status? (Very good/Good/Fair/Poor/Very Poor)